CLINICAL TRIAL: NCT02573207
Title: Recovery of Hibernating Myocardium in End Stage Heart Failure
Acronym: RHIMES-HF
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Intermountain Research and Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pending
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Function After LVAD Implant; Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will collect clinical, echocardiographic, nuclear imaging and hemodynamic data in a group of patients with end stage ischemic cardiomyopathy undergoing left ventricular assist device (LVAD) implantation to investigate the incidence of recovery of myocardial function when supported with LVADs, and to study the association between hibernating myocardium and myocardial recovery in this population.

DETAILED DESCRIPTION:
Clinical, echocardiographic and hemodynamic data will be obtained from the patients' medical records. Assessment of viability will be performed using a Tl-201 Rest-Redistribution Scintigraphy protocol within 2 weeks before LVAD implantation and 2 months after LVAD implant. Recovery of myocardial function will be assessed using available 2D transthoracic echocardiographic images and with the novel imaging modality, Speckle Tracking Echocardiography (STE), in order to provide a regional quantification of the myocardium, in the context of TL-201 results. Transthoracic echocardiograms will be performed 2 weeks prior to the LVAD implant and 1, 2, 3, 4, 6, 9, and 12 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female >= 18 years of age.
2. End stage chronic and dilated ischemic cardiomyopathy requiring LVAD support.
3. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Ischemic cardiomyopathy is defined by a LVEF < 40% and any of the following:

* History of myocardial infarction or revascularization.
* History of angina or chest pain and evidence of scarring in non-invasive imaging studies corresponding to previous myocardial infarction.
* Presence of ≥ 75% stenosis of the left main or proximal left anterior descending artery, or ≥ 75% stenosis of 2 or more epicardial vessels in a patient with unexplained cardiomyopathy.

Exclusion Criteria:

* Pregnant and/or lactating women and women of child bearing potential who are not using acceptable means of contraception. Women of childbearing potential must be using adequate measures of contraception (as determined by the Investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period. Women of childbearing potential must have a negative pregnancy test at screen.
* Patients with acute forms of HF: acute onset of symptoms < 3 months, no left and right ventricular dilation.
* Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>= 18 years old) with end stage ischemic cardiomyopathy receiving a LVAD at the U.T.A.H. Cardiac Transplant Program. We will exclude subjects with acute forms of heart failure and patients with left ventricular ejection fraction (LVEF) < 40% and non-obstructive coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Recovery of Myocardial Function | 2 weeks prior to LVAD implant and 1, 2, 3, 4, 6, 9 and 12 months post LVAD implant
  Recovery of myocardial function assessed continuously, using echocardiographic variables (LVEF, circumferential strain and strain rate, segmental strain and strain rate).

SECONDARY OUTCOMES:
Change in the Proportion of Viable, Hibernating Myocardium and Scar after LVAD Implant | 2 weeks prior to LVAD implant and 2 months post LVAD implant
  Change in the proportion of viable, hibernating myocardium and scar after LVAD implant, measured using Th-201 Rest-Redistribution Viability Study.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah G Kfoury, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Heart Institute, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No